CLINICAL TRIAL: NCT03474627
Title: Sinus Floor Elevation Using Particulate and in Situ Hardening Biphasic Calcium Phosphate Bone Graft Substitutes: A Prospective Histological and Radiological Study
Brief Title: PLGA-coated Biphasic Calcium Phosphate in Sinus Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Full Professor of Oral Surgery and Implant Dentistry, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1452514461215
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Sinus Floor Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-coated HA/TCP particles (Active Comparator): Biphasic hydroxyapatite and beta-tricalcium phosphate bone graft
  Interventions: Device: Non-coated HA/TCP particles
- PLGA-coated HA/TCP particles (Experimental): Biphasic hydroxyapatite and beta-tricalcium phosphate bone graft with PLGA coating
  Interventions: Device: PLGA-coated HA/TCP particles

INTERVENTIONS:
Device: Non-coated HA/TCP particles — Maxillary sinus floor elevation and bone grafting with the use of biphasic hydroxyapatite and beta-tricalcium phosphate bone graft
  Arms: Non-coated HA/TCP particles
Device: PLGA-coated HA/TCP particles — Maxillary sinus floor elevation and bone grafting with the use of biphasic hydroxyapatite and beta-tricalcium phosphate bone graft with PLGA coating
  Arms: PLGA-coated HA/TCP particles

SUMMARY:
The study aims to investigate the radiological and histomorphometric results of the use of PLGA-coated biphasic calcium phosphate granules in sinus floor elevation, to analyze the underlying molecular processes by immunohistochemical staining, and to evaluate the handling of the biomaterial and the in situ hardening properties.

A randomized clinical study is designed to include patients in need of two-stage sinus floor elevation. Patients are assigned to receive either PLGA-coated biphasic calcium phosphate particles (group I) or the equivalent but non-coated particles (group II). CBCT scans are performed before and 6 months after the procedure to assess the bone height gain. At the time of implant placement, bone core biopsies are obtained at the site of implant placement. Histological sections are subjected to histomorphometric and immunohistochemical evaluation of differentiation markers.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients.
* Kennedy class I or II in the upper jaw, from first premolar to second molar.
* Less than 5 mm of residual crestal bone.
* Need for the replacement of teeth with dental implants.

Exclusion Criteria:

* Sinus pathology (sinusitis, mucocele, cysts).
* Smokers.
* Previous long-term (>3 months) use of drugs known to affect bone metabolism, such as bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sinus floor height change | 6 months
  CBCT scans are performed before the sinus floor elevation and 6 months later before implant placement to measure vertical bone height from the crestal bone to the floor of the maxillary sinus.

SECONDARY OUTCOMES:
Area of new mineralized tissue | 6 months
  Histomorphometric quantification of new mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of non-mineralized tissue | 6 months
  Histomorphometric quantification of non-mineralized tissue in a bone biopsy collected 6 months after the grafting procedure
Area of remaining graft particles | 6 months
  Histomorphometric quantification of remaining graft particles in a bone biopsy collected 6 months after the grafting procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Flichy-Fernandez, DDS, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - University of Granada, Granada
  - Universidad de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo-Moreno P, Hernandez-Cortes P, Mesa F, Carranza N, Juodzbalys G, Aguilar M, O'Valle F. Slow resorption of anorganic bovine bone by osteoclasts in maxillary sinus augmentation. Clin Implant Dent Relat Res. 2013 Dec;15(6):858-66. doi: 10.1111/j.1708-8208.2012.00445.x. Epub 2012 Feb 29. PMID 22376122
- [Background] Ortega-Oller I, Del Castillo-Santaella T, Padial-Molina M, Galindo-Moreno P, Jodar-Reyes AB, Peula-Garcia JM. Dual delivery nanosystem for biomolecules. Formulation, characterization, and in vitro release. Colloids Surf B Biointerfaces. 2017 Nov 1;159:586-595. doi: 10.1016/j.colsurfb.2017.08.027. Epub 2017 Aug 24. PMID 28854415
- [Background] Galindo-Moreno P, Avila G, Fernandez-Barbero JE, Aguilar M, Sanchez-Fernandez E, Cutando A, Wang HL. Evaluation of sinus floor elevation using a composite bone graft mixture. Clin Oral Implants Res. 2007 Jun;18(3):376-82. doi: 10.1111/j.1600-0501.2007.01337.x. Epub 2007 Mar 12. PMID 17355356
- [Background] Galindo-Moreno P, de Buitrago JG, Padial-Molina M, Fernandez-Barbero JE, Ata-Ali J, O Valle F. Histopathological comparison of healing after maxillary sinus augmentation using xenograft mixed with autogenous bone versus allograft mixed with autogenous bone. Clin Oral Implants Res. 2018 Feb;29(2):192-201. doi: 10.1111/clr.13098. Epub 2017 Oct 26. PMID 29071736